CLINICAL TRIAL: NCT04560907
Title: Aquablation vs. Holmium Laser Enucleation of the Prostate in the Treatment of Benign Prostatic Hyperplasia in Medium to Large Size Prostates: A Prospective Randomized Trial
Brief Title: Aquablation vs. Holmium Laser Enucleation of the Prostate in the Treatment of Benign Prostatic Hyperplasia in Medium to Large Size Prostates
Acronym: ATHLETE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. med. Gautier Müllhaupt (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Gautier Müllhaupt, Staff member, Sponsor-Investigator, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CantonalHSG
Record Dates: First submitted 2020-09-14; First posted 2020-09-23 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Aquablation

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, non-inferiority clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquablation (Experimental)
  Interventions: Procedure: Aquablation
- HoLEP (Active Comparator)
  Interventions: Procedure: HoLEP

INTERVENTIONS:
Procedure: Aquablation — By means of a high-pressure saline stream, parenchymal tissue of the prostate is removed endoscopically through a heat-free mechanism called hydrodissection. The intervention is supported by live ultrasound guidance and the required depth as well as the angle of the resection is planned out prior to the resection. The bladder is accessed using a 24-Fr hand-piece, which accommodates the scope. The handpiece is supported by an articulating arm attached to the operation table. Once placed in the optimal position, the system automatically adjusts the alignment as necessary.
  Hemostasis is consecutively achieved through diathermy and post procedure, a threeway catheter is inserted and bladder irrigation is initiated.
  Arms: Aquablation
Procedure: HoLEP — This is done endoscopically under general anesthesia the three lobes of the prostate that are cored out intact with the laser are pushed into the bladder before being morcellated by a special instrument inserted through the telescopic camera. A catheter is placed into the bladder to drain the urine while the raw surface heals, then left in place for around 24 hours before being removed on the day of discharge from hospital. Sterile saline fluid is also irrigated into the bladder through the catheter to dilute any blood in the urine and prevent clots from forming.
  Arms: HoLEP

SUMMARY:
Benign prostatic hyperplasia (BPH) is one of the most common diseases in men. As BPH progresses, surgical treatments often become necessary. Holmium enucleation of the prostate (HoLEP) is an established procedure in the surgical treatment of BPH, especially for medium to large prostates. The long learning curve, the length of surgery, and expensive equipment still limit the availability of HoLEP to a few specialized centers.

Recently, a new method for treating BPH called aquablation has become commercially available. This technique uses real-time ultrasound imaging in combination with a robotic high-pressure water jet programmed and guided by the surgeon to resect prostate tissue. A RCT has shown functional results similar to transurethral resection of the prostate (TURP) for small to medium size prostates .

However, so far there are no controlled studies assessing whether Aquablation provides patient reported and functional outcomes that are non-inferior compared to HoLEP in medium size to large prostates (the latter cannot be operated by TURP due to its size limitations).

As aquablation offers some obvious advantages compared to HoLEP regarding learning curve and operation time, the aim of this study is to test whether efficacy and safety of aquablation are non- inferior compared to HoLEP in patients with medium to large size prostates, which would clearly support the use of aquablation and change everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥45 years of age

  * Patient must be a candidate for HoLEP
  * Refractory to medical therapy or patient is not willing to consider (further) medical treatment
  * Patient has a prostate size of at least 50 ml and not more than 150ml, measured by transrectal ultrasound (TRUS)
  * IPSS ≥12
  * QoL≥3
  * Qmax ≤ 15 ml/s with a minimum voided volume ≥ 125 ml or patient in urinary retention
  * Written informed consent

Exclusion Criteria:

* Neurogenic lower urinary tract dysfunction

  * Urethral stenosis
  * Preinterventionally proven adenocarcinoma of the prostate
  * Nickel allergy
  * Not able to complete questionnaires due to cognitive or thought disorders
  * Language skills insufficient for informed consent and / or completion of questionnaires

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-05 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptoms Score (IPSS) | 6 months
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mullhaupt G, Gusewell S, Schmid HP, Zumstein V, Betschart P, Engeler DS, Abt D. Aquablation versus holmium laser enucleation of the prostate in the treatment of benign prostatic hyperplasia in medium-to-large-sized prostates (ATHLETE): protocol of a prospective randomised trial. BMJ Open. 2021 May 3;11(5):e046973. doi: 10.1136/bmjopen-2020-046973. PMID 33941632